CLINICAL TRIAL: NCT02845193
Title: Effect of A Novel (Modified Grayson) Technique for Nasoalveolar Molding and Taping on Parents' Satisfaction and Short Term Treatment Outcomes in Infants With Unilateral Complete Cleft Lip and Palate: A Randomized Controlled Trial
Brief Title: Effect of Novel Nasoalveolar Molding Techniques on Parents' Satisfaction and Short Term Treatment Outcomes in Unilateral Cleft Lip and Palate Infants: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abd El-Ghafour, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-2016-07-172
Record Dates: First submitted 2016-07-19; First posted 2016-07-27 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Modified Nasoalveolar molding group (Experimental): This group will receive nasoalveolar molding appliance in addition to taping for 3 Months with follow-up every 2 weeks.
  Interventions: Device: Modified Nasoalveolar molding
- Taping group (Experimental): Tape will be used alone in this group on the upper lip segments for 3 months with follow-up every 2 weeks.
  Interventions: Device: Taping
- Control group (No Intervention): This group will not receive any treatment.
- CAD/NAM group (Experimental): Computer Aided Designed Nasoalveolar molding and 3D printed.
  Interventions: Device: CAD/NAM

INTERVENTIONS:
Device: Modified Nasoalveolar molding — Infants will receive this appliance which is a maxillary plate with nasal stent in addition to taping on the upper lip (taping is routine step in Grayson's nasoalveolar molding technique).
  Arms: Modified Nasoalveolar molding group
Device: Taping — Infants will receive a tape only on the upper lip segments to mold it to touch each other.
  Arms: Taping group
Device: CAD/NAM — computer aided design NAM
  Arms: CAD/NAM group

SUMMARY:
The aim of this trial is to figure out the efficiency of modified Grayson NAM on parents' satisfaction, nasal esthetics, interlabial gap and maxillary arch changes. NAM might improve and facilitate the surgical procedure after lip closure. This might decrease the need of further interventions to improve esthetics and function of CLP patients. This trial will help the patients and practitioners in taking the decision of inclusion of NAM in the CLP treatment protocol as a mandatory step or skip a useless procedure with all of its burden.

DETAILED DESCRIPTION:
In this randomized trial, 4 groups will be included. The first group will receive a modified nasoalveolar molding appliance in addition to taping. In the second group, the patient will receive the CAD/NAM. the third group is tape only, while the fourth group remain untreated. the follow-up period will be 3 months till surgical lip closure. the assessment will be through a questionnaire for the parents' satisfaction outcome, photographs for nasal esthetics and interlabial gap outcome and maxillary models for the maxillary dimension change outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with age range from 7 - 30 days.
2. Unilateral complete cleft lip and alveolus.
3. Presence of unilateral cleft palate.
4. Medically free subjects.
5. Both males and females.

Exclusion Criteria:

1. Patients older than 30 days.
2. Syndromic patients with other defects in addition to cleft lip and palate.
3. Patients with bilateral cleft lip and palate.
4. Incomplete Cleft lip.
5. Medically compromised patients.

Ages: 7 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Parents' satisfaction | 3 months
  It will be assessed using Questionnaire.

SECONDARY OUTCOMES:
Nasal Esthetics: a- Nostril height | 3 months
  It will be measured in mm by Digital ruler on the images using a software.
Nasal Esthetics: b- Nostril width | 3 months
  It will be measured in mm by Digital ruler on the images using a software.
Nasal Esthetics: c- Nasal sill height | 3 months
  It will be measured in mm by Digital ruler on the images using a software.
Nasal Esthetics: d- Nostril area | 3 months
  It will be measured on the images in mm 2 (square) using a software measuring area.
Interlabial gap | 3 months
  It will be measured in mm by Digital ruler on the images using a software.
Maxillary Arch Dimension | 3 months
  It will be measured as distances in mm between landmarks identified on the dental models assessing the anterioposterior, transverse and vertical changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Abd El-Ghafour M, Aboulhassan MA, El-Beialy AR, Fayed MMS, Eid FHK, Emara D, El-Gendi M. Does Presurgical Taping Change Nose and Lip Aesthetics in Infants with Unilateral Cleft Lip and Palate? A Randomized Controlled Trial. Plast Reconstr Surg. 2022 Dec 1;150(6):1300e-1313e. doi: 10.1097/PRS.0000000000009738. Epub 2022 Sep 20. PMID 36126199